CLINICAL TRIAL: NCT01510847
Title: The Effect of 90-day Oral Testosterone Therapy in Chinese Males With Type 2 Diabetes: OTEST
Brief Title: The Effect of 90-day Oral Testosterone Therapy in Chinese Males With Type 2 Diabetes (T2DM)
Acronym: OTEST
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Unable to reach the target recruitment within timeline
Sponsor: Singapore Clinical Research Institute (Other)
Collaborators: Singapore General Hospital (Other); Duke-NUS Graduate Medical School (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: OTEST/SCRI; DUKE-NUS-TIDR/2010/0001 (Other: Singapore Clinical Research Institute PL/DUKE-NUS Singapore)
Record Dates: First submitted 2012-01-04; First posted 2012-01-18 (Estimated); Last update posted 2016-01-06 (Estimated); Status verified 2016-01

CONDITIONS: Assess the Effects of a the 90-day Oral TS Study Regimen on PSA, IPSS, Haemoglobin and Haematocrit, and to Assess Adverse and Serious Adverse Events.

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Oral Testosterone Therapy (Other): 90 day oral testosterone therapy
  Interventions: Drug: Andriol Testocaps

INTERVENTIONS:
Drug: Andriol Testocaps — Oral, 40mg, Twice a day, 30days

SUMMARY:
The study hypothesis is that treatment with oral Testosterone according to the study regimen will improve glycemic control in T2DM Chinese males in Singapore as indicated by a reduction in HbA1c levels at study day 90.

DETAILED DESCRIPTION:
This is a single arm open label clinical study in Chinese men of 45 to 75 years of age with Type 2 Diabetes. Subjects will be recruited from participating family medicine clinics with the FMRN and followed for 90-days. All subjects will continue on pre-study treatment regimens and medications as clinically indicated throughout the 90-day study period. Missed doses of study drug can be made up within the same day. With the exceptions of study drug and diabetic medications, changes in other medications will be permitted. The primary aim is to assess the effects of oral Testosterone on change in HbA1c levels in the Chinese males with a diagnosis of T2DM over a 90-day study period.

Subjects enrolled in the study will take two 40mg capsules of oral testosterone in the morning and two 40mg capsules in the evening with meals on both occasions on each day. This daily dosage is consistent with the recommended dosage for subjects being treated for hypogonadism.

Primary objective:

- The primary aim is to assess the effect of oral Testosterone on percent change in HbA1c in T2DM Chinese males in Singapore over a 90-day study period.

Secondary objectives:

- The secondary aim is to assess the effects of site, eugonadism and hypogonadism, and the prognostic relevance of baseline levels of HbA1c, total testosterone, PSA, IPSS, haemoglobin and haematocrit on 90-day change and percent change from baseline in HbA1c under the study Testosterone regimen.

All subjects must satisfy ALL of the following criteria at study entry:

* Subject is a Chinese male
* Subject is 45 to 75 years old
* Subject has T2DM with no change in type/dose of diabetic medication in the last 3 months
* Subject's Haemoglobin level is between 13.5 - 18g/dl
* Subject's Haematocrit level is 40 - 54%
* Subject's Albumin level is between 3.5 - 5.0 g/dL
* Subject's Alanine transaminase (ALT) level is up to 36 U/L
* Subject's Aspartate transaminase (AST) level is < 41 U/L
* Subject's Alkaline phosphatase (ALP) level is < 130 U/L
* Subject's Creatinine(up to 60 years) level is between 0.57 - 1.36 mg/dL
* Subject's Creatinine(> 60 years) level is between 0.68 - 1.48 mg/dL
* Subject's Sodium(13 to 65 years) level is between 136 - 145 mmol/L
* Subject's Sodium(> 65 years) level is between 132 - 146 mmol/L
* Subject's Potassium (up to 59 years) level is between 3.3 - 5.1 mmol/L
* Subject's Potassium (> 59 years) level is between 3.7 - 5.4 mmol/L
* Subject's PSA (Prostate Specific Antigen) level is ≤ 4ug/L
* Subject's Total Testosterone level is between 8.4 - 28.7 nmol/L
* Satisfactory haematological or biochemical functions tests only - these tests should be carried out during the screening period prior to enrolment. Patient with mild laboratory abnormalities can be included at the discretion by the site/co-investigator, and after approval by Co-ordinating Principal Investigator
* Written Informed Consent is obtained
* Subject is willing to comply with study procedures and is able to return to the clinic for scheduled visits

All subjects must NOT have any of the following criteria at study entry:

* Subject's HbA1C level is > 9%.
* Subject is on insulin therapy
* Subject has history of recurrent hypoglycaemia
* Subject has history of malignancy (except skin cancer) during last 5 years
* Subject has received treatment for endocrinopathy within the last 3 months (except diabetes)
* Subject has history of adverse drug reaction to testosterone
* Subject has received testosterone replacement within the last 3 months
* Subject is currently receiving warfarin, steroids, cyclosporine or thyroxine
* Subject has history of Myocardial Infarction
* Subject has history of Angina
* Subject has heart failure which causes at least slight limitation of physical activity. Subject is comfortable at rest, but ordinary physical activity results in fatigue, palpitation or dyspnea
* Subject has history of Deep Vein Thrombosis or Stroke
* Subject has history of prostate cancer
* Subject has history of chronic kidney disease , Stage 3 or worse
* Subject has life expectancy of less than 1 year
* Subject has enlarged prostate per digital rectal examination
* Subject's International Prostate Symptom Score (IPSS) is greater than 20

Blood samples will be drawn during the study period:

* 16 types of blood samples at Baseline, Month 1 and Month 3 Visits.
* HbA1c, Haemoglobin, Haematocrit, Albumin, ALT, AST, ALP,Creatinine,PSA, Total Testosterone, Total Cholesterol,HDL, LDL, Triglycerides, Sodium,Potassium

ELIGIBILITY:
Inclusion Criteria:

* Subject is a Chinese male
* Subject is 45 to 75 years old
* Subject has T2DM with no change in type/dose of diabetic medication in the last 3 months
* Subject 's Haemoglobin level is between 13.5 - 18g/dl
* Subject's Haematocrit level is 40 - 54%
* Subject's Albumin level is between 3.5 - 5.0 g/dL
* Subject's Alanine transaminase (ALT) level is up to 36 U/L
* Subject's Aspartate transaminase (AST) level is < 41 U/L
* Subject's Alkaline phosphatase (ALP) level is < 130 U/L
* Subject's Creatinine (up to 60 years) level is between 0.57 - 1.36 mg/dL
* Subject's Creatinine (> 60 years) level is between 0.68 - 1.48 mg/dL
* Subject's Sodium (13 to 65 years) level is between 136 - 145 mmol/L
* Subject's Sodium ( > 65 years) level is between 132 - 146 mmol/L
* Subject's Potassium ( up to 59 years) level is between 3.3 - 5.1 mmol/L
* Subject's Potassium ( > 59 years) level is between 3.7 - 5.4 mmol/L
* Subject's PSA (Prostate Specific Antigen) level is ≤ 4ug/L
* Subject's Total Testosterone level is between 8.4 - 28.7 nmol/L
* Satisfactory haematological or biochemical functions tests only - these tests should be carried out during the screening period prior to enrolment. Patient with mild laboratory abnormalities can be included at the discretion by the site/co-investigator, and after approval by Co-ordinating Principal Investigator
* Written Informed Consent is obtained
* Subject is willing to comply with study procedures and is able to return to the clinic for scheduled visits

Exclusion Criteria:

* Subject's HbA1C level is > 9%.
* Subject is on insulin therapy
* Subject has history of recurrent hypoglycaemia
* Subject has history of malignancy (except skin cancer) during last 5 years
* Subject has received treatment for endocrinopathy within the last 3 months (except diabetes)
* Subject has history of adverse drug reaction to testosterone
* Subject has received testosterone replacement within the last 3 months
* Subject is currently receiving warfarin, steroids, cyclosporine or thyroxine
* Subject has history of Myocardial Infarction
* Subject has history of Angina
* Subject has heart failure which causes at least slight limitation of physical activity. Subject is comfortable at rest, but ordinary physical activity results in fatigue, palpitation or dyspnea
* Subject has history of Deep Vein Thrombosis or Stroke
* Subject has history of prostate cancer
* Subject has history of chronic kidney disease , Stage 3 or worse
* Subject has life expectancy of less than 1 year
* Subject has enlarged prostate per digital rectal examination
* Subject's International Prostate Symptom Score (IPSS) is greater than 20

Ages: 45 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2011-10; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
The Effect of 90-day Oral Testosterone Therapy in Chinese Males with Type 2 Diabetes (T2DM): OTeST | 90 Day Study Period
  The primary aim is to assess the effect of oral Testosterone Supplementation on percent change in HbA1c in Type 2 Diabetes Mellitus Chinese males in Singapore over a 90-day study period.

SECONDARY OUTCOMES:
The Effect of 90-day Oral Testosterone Therapy in Chinese Males with Type 2 Diabetes (T2DM): OTeST | 90 day study period
  The secondary aim is to assess the effects of site, eugonadism and hypogonadism, and the prognostic relevance of baseline levels of HbA1c, total testosterone, PSA, IPSS, haemoglobin and haematocrit on 90-day change and percent change from baseline in HbA1c under the study Testosterone Supplementation regimen.

CONTACTS AND LOCATIONS:
Overall Officials: Sam Lim, MBBS, Principal Investigator — Singapore Clinical Research Institute Pte Lte
Locations (12):
- Singapore (12):
  - Camry Medical Centre, Singapore, Singapore
  - Frontier Medical Associates (Ubi) Pte Ltd, Singapore, Singapore
  - Everhealth Medical Centre, Singapore, Singapore
  - Frontier Medical Associates (Buangkok Cresent) Pte Ltd, Singapore, Singapore
  - Frontier Medical Associates (AMK) Pte Ltd, Singapore, Singapore
  - EJ Tan Clinic & Surgery, Singapore, Singapore
  - Everhealth Family Clinic & Surgery, Singapore, Singapore
  - Bukit Batok Medical Clinic, Singapore, Singapore
  - Princeton Family Clinic Pte Ltd, Singapore, Singapore
  - The Edinburgh Clinic, Singapore, Singapore
  - Frontier Medical Associates (Woodlands) Pte Ltd, Singapore, Singapore
  - Frontier Medical Associates (Yishun) Pte Ltd, Singapore, Singapore